CLINICAL TRIAL: NCT01569204
Title: Targeted BEACOPP Variants in Patients With Newly Diagnosed Advanced Classical Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. Peter Borchmann, Prof., University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Targeted BEACOPP
Record Dates: First submitted 2012-04-02; First posted 2012-04-03 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Etoposide; Cyclophosphamide; Doxorubicin; Prednisone; Procarbazine; Dexamethasone; Dacarbazine; Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BrECAPP (Active Comparator): modified BEACOPP by omitting Bleomycin and adding Brentuximab Vedotin
  Interventions: Drug: Etoposide; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone; Drug: Procarbazine; Drug: Brentuximab Vedotin
- BrECADD (Active Comparator): modified BEACOPP by omitting Bleomycin, Procarbazine and Prednisone and adding Brentuximab Vedotin, Dacarbazine and Dexamethasone
  Interventions: Drug: Etoposide; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Dexamethasone; Drug: Dacarbazine; Drug: Brentuximab Vedotin

INTERVENTIONS:
Drug: Etoposide
Drug: Cyclophosphamide
Drug: Doxorubicin
Drug: Prednisone
  Arms: BrECAPP
Drug: Procarbazine
  Arms: BrECAPP
Drug: Dexamethasone
  Arms: BrECADD
Drug: Dacarbazine
  Arms: BrECADD
Drug: Brentuximab Vedotin

SUMMARY:
The Purpose of this trial is:

* to determine complete response rate (CRR) after six cycles of chemotherapy
* to determine complete remission rate (CR/CRr) as final treatment outcome after completion of treatment

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven classical Hodgkin lymphoma
* First diagnosis, no previous treatment, age: 18-60 years
* Stage IIB with large mediastinal mass and/or extranodal lesions, stage III or IV disease

Exclusion Criteria:

* Composite lymphoma or nodular lymphocyte- predominant Hodgkin lymphoma (NLPHL)
* Previous malignancy
* Prior chemotherapy or radiation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Response rate (RR) after six cycles of chemotherapy | 18 weeks
Complete remission rate (CR/CRr) as final treatment outcome after completion of treatment | 18 weeks

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 2 years
Overall survival (OS) | 2 years
Adverse event rate | 2 years
Dose reduction rate | 18 weeks
Relative dose intensity | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Borchmann, Prof., Principal Investigator — University of Cologne, German Hodgkin Study Group
Locations (1):
- 1st Dept. of Medicine, Cologne University Hospital, Cologne, Germany

REFERENCES:
- See also: Homepage GHSG — http://www.ghsg.org